CLINICAL TRIAL: NCT07300189
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of TLC-1180 in Healthy Subjects and an Open-Label Assessment of the Relative Bioavailability of, and Effect of Food on, a Tablet Formulation of TLC-1180
Brief Title: A Study to Evaluate Single and Multiple Doses of TLC-1180 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OrsoBio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1180-CL-101
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Solution (Experimental): Oral solution of TLC-1180
  Interventions: Drug: TLC-1180 Oral Solution; Other: Placebo Oral Solution
- Tablet (Experimental): Tablet formulation of TLC-1180
  Interventions: Drug: TLC-1180 Tablet; Other: Placebo Tablet

INTERVENTIONS:
Drug: TLC-1180 Oral Solution — Oral solution of TLC-1180
  Arms: Oral Solution
Drug: TLC-1180 Tablet — Tablet formulation of TLC-1180
  Arms: Tablet
Other: Placebo Oral Solution — Placebo-to-match oral solution TLC-1180
  Arms: Oral Solution
Other: Placebo Tablet — Placebo-to-match tablet formulation of TLC-1180
  Arms: Tablet

SUMMARY:
This phase 1 study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of TLC-1180 after single- and multiple-ascending doses in healthy subjects.

DETAILED DESCRIPTION:
The primary objectives are to assess the safety, tolerability, and plasma PK of TLC-1180 in healthy subjects. The exploratory objective is to evaluate the PD of TLC-1180 in healthy subjects. This study is comprised of four parts: Part A (single-ascending dose), Part B (multiple-ascending dose), optional Part C (adaptive single- and/or multiple-ascending dose), and Part D (relative bioavailability of a tablet formulation of TLC-1180). Up to 72, 100, 100, and 8 healthy subjects will be recruited in Parts A, B, C, and D, respectively. The effect of food on TLC-1180 PK will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy male or female subject between 18 and 55 years of age, inclusive
* Body mass index from 19 to 35 kg/m2, inclusive
* Estimated glomerular filtration rate ≥ 80 mL/min
* Normal liver biochemistry tests
* Screening laboratory evaluations (hematology, chemistry, and urinalysis) must fall within the normal range of the local laboratory's reference ranges unless the results have been determined by the investigator to have no clinical significance
* Subject must have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the investigator
* Females of childbearing potential must have a negative pregnancy test at Screening and clinic admission
* Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception
* Must, in the opinion of the investigator, be in good health based upon medical history and physical examination, including vital signs

Exclusion Criteria:

* Pregnant or lactating subjects
* Subjects who have any serious or active medical or psychiatric illness (including depression) that, in the opinion of the investigator, would interfere with the subject's treatment, assessment, or compliance with the protocol
* Subjects who have received any investigational compound within 30 days or 5 half-lives, whichever is longer, prior to study drug dosing
* Current alcohol abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* Current substance abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* A positive test result for human immunodeficiency virus (HIV-1) antibody, hepatitis B (HBV) surface antigen, or hepatitis C (HCV) antibody
* Subjects who have taken any prescription medications or over-the-counter medications, including herbal products, within 28 days prior to start of study drug dosing, with the exception of vitamins, acetaminophen (paracetamol), ibuprofen, and/or hormonal contraceptive medications
* Subjects who have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to Screening or expected to receive these agents during the study (e.g., corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies)
* Medical history of serious skin disease in the opinion of the investigator, such as but not limited to rash, food allergy, eczema, psoriasis, or urticaria
* Medical history of drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity)
* Presence or history of cardiovascular disease, including significant cardiovascular disease (including a history of myocardial infarction based on ECG and/or clinical history), history of cardiac conduction abnormalities (including any history of ventricular tachycardia), congestive heart failure, cardiomyopathy with left ventricular ejection fraction < 40%, a family history of Long QT Syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years
* Syncope, palpitations, or unexplained dizziness
* Implanted defibrillator or pacemaker
* Medical history of liver disease, including but not limited to alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency)
* History of rhabdomyolysis
* Severe peptic ulcer disease, gastroesophageal reflux disease, or other gastric acid hypersecretory conditions
* History of medical or surgical treatment that permanently alters intestinal absorption (e.g., gastric or intestinal surgery)
* Subjects who have received vaccination for COVID-19 within 14 days of Admission

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of TLC-1180 treatment-emergent adverse events | Through study completion: Day 57 (Parts A, C); Day 28 (Parts B, C); Day 39 (Part D) of the study
  Adverse events (AEs) - severity of the AEs will be graded using the Common Terminology Criteria for AE (CTCAE) (v5.0). The relationship between AEs and the study drug will be indicated as related or not related.
PK of TLC-1180 AUC | Through study completion: Day 57 (Parts A, C); Day 28 (Parts B, C); Day 39 (Part D) of the study
  Area under the concentration-time curve
PK of TLC-1180 Cmax | Through study completion: Day 57 (Parts A, C); Day 28 (Parts B, C); Day 39 (Part D) of the study
  Maximum plasma concentration
PK of TLC-1180 tmax | Through study completion: Day 57 (Parts A, C); Day 28 (Parts B, C); Day 39 (Part D) of the study
  Time to reach Cmax
PK of TLC-1180 t1/2 | Through study completion: Day 57 (Parts A, C); Day 28 (Parts B, C); Day 39 (Part D) of the study
  Half-life
PK of TLC-1180 CL/F | Through study completion: Day 57 (Parts A, C); Day 28 (Parts B, C); Day 39 (Part D) of the study
  Apparent clearance, calculated as dose/AUC0-inf

CONTACTS AND LOCATIONS:
Locations (1):
- OrsoBio Research Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No